CLINICAL TRIAL: NCT03268902
Title: Early Life Interventions for Childhood Growth and Development In Tanzania
Acronym: ELICIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Haydom Lutheran Hospital (Other)
Collaborators: University of Virginia (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19465
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Malnutrition; Stunting; Cognitive Development; Enteric Pathogens
MeSH Terms: conditions — Malnutrition; Growth Disorders | interventions — nitazoxanide; Niacinamide

STUDY DESIGN:
Intervention Model Description: Each intervention will be assigned independently. Intervention domains will be randomized separately on an individual basis. This will provide 4 different combinations of interventions: 1). Nicotinamide, azithromycin and nitazoxanide 2). Azithromycin and nitazoxanide 3). Nicotinamide only 4). No active treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and investigators will be blinded to the treatments allocated to each participant. The members of the DSMB will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Nicotinamide and Antimicrobials (Experimental): Nicotinamide Azithromycin Oral Liquid Product Nitazoxanide Oral Suspension
  Interventions: Drug: Azithromycin Oral Liquid Product; Drug: Nitazoxanide Oral Suspension; Dietary Supplement: Nicotinamide
- Antimicrobials only (Experimental): Placebo Azithromycin Oral Liquid Product Nitazoxanide Oral Suspension
  Interventions: Drug: Azithromycin Oral Liquid Product; Drug: Nitazoxanide Oral Suspension; Drug: Placebos
- Nicotinamide only (Experimental): Nicotinamide Placebo Placebo
  Interventions: Dietary Supplement: Nicotinamide; Drug: Placebos
- No active treatment (Placebo Comparator): Placebo Placebo Placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Azithromycin Oral Liquid Product — Azithromycin 20 mg/kg administered by study personnel at 6, 9, 12 and 15 months
  Other Names: Throza DPS
  Arms: Antimicrobials only; Nicotinamide and Antimicrobials
Drug: Nitazoxanide Oral Suspension — Nitazoxanide 100 mg given twice daily for 3 days at 12 and 15 months
  Other Names: Alinia
  Arms: Antimicrobials only; Nicotinamide and Antimicrobials
Dietary Supplement: Nicotinamide — Mothers in the nicotinamide arm will be given nicotinamide 250 mg daily from delivery through 6 months post-partum in capsule form.
  Children in the nicotinamide arm will be given 100 mg/d in powder form between 6 and 18 months of age
  Other Names: Vitamin B3
  Arms: Nicotinamide and Antimicrobials; Nicotinamide only
Drug: Placebos — Contain inert excipients only. Azithromycin placebo 20 mg/kg administered by study personnel at 6, 9, 12 and 15 months. Nitazoxanide placebo 100 mg given twice daily for 3 days at 12 and 15 months.
  Mothers in the nicotinamide placebo arm will be given placebo 250 mg daily from delivery through 6 months post-partum in capsule form.
  Children in the nicotinamide placebo arm will be given 100 mg/d of placebo in powder form between 6 and 18 months of age
  Arms: Antimicrobials only; Nicotinamide only; No active treatment

SUMMARY:
This study aims to assess growth and cognitive effects of treatment with azithromycin and nitazoxanide and/or nicotinamide (vitamin B3) supplementation nicotinamide.

DETAILED DESCRIPTION:
Children living in rural sub-Saharan Africa experience massive challenges to child thriving, with poor linear growth and delays in child development. In a cohort of 211 children living in the rural Haydom area of Tanzania (participating in the Interactions of Malnutrition & Enteric Infections: Consequences for Child Health and Development "MAL-ED" Study), 70.6% had stunted growth at 18 months. This rate of moderate and severe stunting (length-for-age z-score [HAZ] <-2 standard deviations) was the highest of the 8 study sites in MAL-ED.

This enormous deficit is likely associated with high rates of enteric infections with Campylobacter, E. coli pathotypes, Cryptosporidium, and Giardia, organisms susceptible to azithromycin and/or nitazoxanide. Infections such as these occur frequently in developing areas and are often associated with environmental enteropathy, including ongoing enteric inflammation and loss of enterocyte integrity, leading to possible bacterial translocation and poorer absorption of ingested nutrients. The consequences of these infections, enteric dysfunction and poor nutrient absorption frequently include growth stunting, learning delays, and an overall loss of human capital.

Emerging evidence suggests a potential role for the tryptophan-niacin pathway (including the end-product nicotinamide, an isoform of vitamin B3) in decreasing mucosal inflammation and affecting enteral microbiota. At the Tanzania site of MAL-ED, serum levels of tryptophan were related to subsequent linear growth, further suggesting importance of the tryptophan-niacin pathway. What is not clear is whether early childhood growth and development could be improved by targeting enteric infection and the tryptophan-niacin pathway by 1) delivering antibiotics against specific bacteria and/or 2) providing vitamin B3 as nicotinamide/niacinamide.

The main analysis will be intention-to-treat but a secondary analysis will be per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age ≥18
2. Infant ≤ 14 days

Exclusion Criteria:

1. Maternal inability to adhere to protocol
2. Multiple gestation
3. Severe illness (significant birth defect, hospitalization, severe neonatal illness)
4. Birth weight <1500 g
5. Lack of breastfeeding at enrollment (and lack of intention to continue breastfeeding at time of enrollment).

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1188 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Height-for-age z-score (HAZ) at 18 months | 18 months

SECONDARY OUTCOMES:
Weight-for-age z-score (WAZ) at 18 months | 18 months
Head circumference-for-age z-score (HCAZ) at 18 months | 18 months
Stunting | 18 months
  HAZ <-2
All cause mortality | 0-18 months
Hospitalization | 0-18 months
Childhood illness | 0-18 months
  Incidence of diarrhea, lower respiratory infection and febrile illness
Anemia | 12 and 18 months
  Moderate to severe anemia by WHO definition for age and altitude
Enteropathogen burden | 6, 6.5, 12, 12.5, 18 months
Microbiota composition | 6, 6.5, 12, 18 months
  Composition of intestinal microbiome
Stool myeloperoxidase concentration | 6, 12, 18 months
  Stool myeloperoxidase ELISA
C-reactive protein concentration in serum | 12 and 18 months
  High-sensitivity CRP concentration
Insulin-like growth factor 1 concentration in serum | 12 and 18 months
Collagen X concentration in serum | 12 and 18 months
Tryptophan-kynurenine ratio | 12 and 18 months
  Ratio of tryptophan concentration to kynurenine concentration in metabolomic testing
Niacin and nicotinamide metabolite concentration | 6, 12, 18 months
  Concentration of downstream metabolites of niacin and nicotinamide as tested by metabolomic analysis
Small intestinal bacterial overgrowth | 6, 12 and 18 months
  Prevalence of SIBO as tested via exhaled hydrogen
Malawi Developmental Assessment Tool score | 18 months
  The MDAT is a measure of child cognitive development

CONTACTS AND LOCATIONS:
Overall Officials: Estomih Mduma, Principal Investigator — Haydom Lutheran Hospital
Locations (1):
- Haydom Lutheran Hospital, Haydom, Manyara Region, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeBoer MD, Elwood SE, Guga G, Jatosh S, Scharf RJ, Liu J, Rogawski McQuade ET, Mduma ER, Houpt E, Platts-Mills JA. Enteric pathogen carriage in early childhood is associated with elevated CRP, lower IGF-1 and linear growth deficits: the ELICIT study in rural Tanzania. BMJ Glob Health. 2025 Nov 12;10(11):e018454. doi: 10.1136/bmjgh-2024-018454. PMID 41232946
- [Derived] Parpia T, Elwood S, Rogawski McQuade ET, Svensen E, Wanjuhi A, Jatosh S, Bayo E, Hhando E, Houpt ER, Mduma E, DeBoer MD, Scharf RJ, Platts-Mills JA. Growth and Cognitive Development in Tanzanian Children are Associated with Timing of Birth in Relation to Seasonal Malnutrition. J Pediatr. 2024 Dec;275:114202. doi: 10.1016/j.jpeds.2024.114202. Epub 2024 Jul 19. PMID 39032770
- [Derived] DeBoer MD, Elwood SE, Platts-Mills JA, McDermid JM, Scharf RJ, Rogawski McQuade ET, Jatosh S, Houpt ER, Mduma E. Association of Circulating Biomarkers with Growth and Cognitive Development in Rural Tanzania: A Secondary Analysis of the Early Life Interventions in Childhood Growth and Development In Tanzania (ELICIT) Study. J Nutr. 2023 May;153(5):1453-1460. doi: 10.1016/j.tjnut.2023.03.020. Epub 2023 Mar 22. PMID 36963502
- [Derived] DeBoer MD, Platts-Mills JA, Elwood SE, Scharf RJ, McDermid JM, Wanjuhi AW, Jatosh S, Katengu S, Parpia TC, Rogawski McQuade ET, Gratz J, Svensen E, Swann JR, Donowitz JR, Mdoe P, Kivuyo S, Houpt ER, Mduma E. Effect of scheduled antimicrobial and nicotinamide treatment on linear growth in children in rural Tanzania: A factorial randomized, double-blind, placebo-controlled trial. PLoS Med. 2021 Sep 28;18(9):e1003617. doi: 10.1371/journal.pmed.1003617. eCollection 2021 Sep. PMID 34582462
- [Derived] DeBoer MD, Platts-Mills JA, Scharf RJ, McDermid JM, Wanjuhi AW, Gratz J, Svensen E, Swann JR, Donowitz JR, Jatosh S, Houpt ER, Mduma E. Early Life Interventions for Childhood Growth and Development in Tanzania (ELICIT): a protocol for a randomised factorial, double-blind, placebo-controlled trial of azithromycin, nitazoxanide and nicotinamide. BMJ Open. 2018 Jul 7;8(7):e021817. doi: 10.1136/bmjopen-2018-021817. PMID 29982218

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT03268902/SAP_002.pdf